CLINICAL TRIAL: NCT06768970
Title: A Decentralized Clinical Trial to Investigate the Effect of Daily Cardio Capsules (US FDA NDI) Supplementation on Improved Sleep in Healthy, Urban-Dwelling Adult Participants
Brief Title: Investigating the Effect of Daily CARDIO® Capsules Supplementation on Improved Sleep in Healthy, Urban-Dwelling Adults
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hofseth Biocare ASA (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: OmeGo-Sleep-001
Record Dates: First submitted 2024-03-01; First posted 2025-01-10 (Actual); Last update posted 2025-01-10 (Actual); Status verified 2025-01

CONDITIONS: Sleep; Pollution; Exposure; Cough
Keywords: salmon oil; sleep quality; environmental pollution; decentralized; virtual platform; clinical trial
MeSH Terms: conditions — Cough; Sleep Initiation and Maintenance Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- CARDIO® Capsules (2.0 g) (Experimental): The study intervention entails CARDIO® salmon oil supplementation, a nutritional product containing a full spectrum of omega fatty acids. Participants allocated to the 2g/d arm will receive two capsules daily as their dosage regimen.
  Interventions: Dietary Supplement: CARDIO® salmon oil
- CARDIO® Capsules (4.0 g) (Experimental): The study intervention entails CARDIO® salmon oil supplementation, a nutritional product containing a full spectrum of omega fatty acids. Participants allocated to the 4g/d arm will receive four capsules daily as their dosage regimen.
  Interventions: Dietary Supplement: CARDIO® salmon oil

INTERVENTIONS:
Dietary Supplement: CARDIO® salmon oil — CARDIO® is a natural salmon oil manufactured from the enzymatic hydrolysis of Norwegian Atlantic salmon. Salmon capsules contain a full spectrum omega- and non-omega marine fatty acids with naturally occurring astaxanthin.
  Other Names: OmeGo

SUMMARY:
This study aims to explore the impact of supplementation with CARDIO® whole salmon oil capsules on healthy adult participants with sleep disruption related to particulate matter pollution. The trial will employ a decentralized approach enabled by modern technology and wearables to measure sleep quantity and quality. Validated patient reported outcome (PRO) measures will be employed to measure the impact on cough and the subjective assessment of sleep quality and wellbeing. After a two week run-in period, subjects will be randomized to OmeGo at either 2g or 4g daily for 8 weeks. Final assessment will be at week 10.

DETAILED DESCRIPTION:
This study aims to explore the impact of a nutritional supplement, CARDIO® salmon oil, on sleep quality and cough among adults residing in urban areas with air quality index / AQI 50 or higher. The trial will employ a decentralized approach enabled by modern technology and wearables. The co-primary endpoint is sleep quality, as measured by wearable device, and impact on cough measured via patient reported outcomes (visual analogue scale / VAS). Secondary endpoints will measure subjective change in sleep via participant-reported VAS and voluntary nasal swabs will be taken in up to 40 participants to assess change in gene expression of relevant cytokines and chemokines. Due to the exploratory nature of this study a placebo arm is not being employed, rather participants will be randomized to CARDIO® at either 2g or 4g daily for 8 weeks following a two-week run-in period where baseline sleep metrics will be recorded by wearable device and the Epworth Sleepiness Scale to measure daytime sleepiness. Final assessment will be undertaken in week 10.

ELIGIBILITY:
Inclusion Criteria:

* Age

  * Participants must be between 18 and 70 years of age.
* Technological access

  * Must possess the ability to access and operate a mobile or web-based device manufactured after 2008.
* Sleep disturbed by coughing resulting in daytime tiredness
* Level of cough burden over previous 24 hours self-scored at ≥40mm on the 0mm ("no cough problems") to 100mm ("most troublesome cough") cough level on visual analog scale (VAS) at screening and baseline
* Wearable Technology

  * Ownership of a wearable device that collects and records time spent in different sleep stages (e.g., REM, Deep, Light, Awake), such as an Apple Watch, Whoop, Google Fit, Fitbit, Garmin, or Oura ring device.

Exclusion Criteria:

Medication Restrictions:

* Use of neuromodulatory therapy (latter including gabapentin, pregabalin, morphine and amitriptyline).
* Current use of ACE (angiotensin converting enzyme) inhibitors or have taken an ACE inhibitor within 3 months of screening.

Pregnant or lactating women

Smoking Status:

● Individuals who are smokers or have smoked within the past 12 months.

Sleep Aid Limitations:

● Use of prescription or over-the-counter sleep aids, including both wellness and prescribed medications.

Sleep Disorder Diagnosis:

* The presence of diagnosed sleep disorders. Alcohol
* Alcohol abuse (4 drinks per day for women and more than 12 per week and 5 or more per day for men or more than 15 drinks per week) or substance use disorder.

Supplement Constraints:

● Use of fish oil, other marine oils (including algal or krill) and omega supplements is not allowed for the duration of the study, with a prerequisite of abstaining from these supplements for at least 3 months prior to participation.

Allergic to fish Epworth Sleepiness Scale score of ≥16

• Any participant with a score of ≥16 will be advised to seek medical attention before entering the study to ensure that they have no undiagnosed medical conditions. If they are deemed medically fit and well they will be able to continue in the study.

Lifestyle Considerations No change in dietary habits, caffeine or alcohol intake or activities of daily living.

No shift work involving night shifts No change in use of vitamins and minerals

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 131 (Actual)
Dates: Start 2024-05-14 (Actual); Primary Completion 2024-11-15 (Actual); Study Completion 2025-01-05 (Actual)

PRIMARY OUTCOMES:
The impact of OmeGo capsules on sleep quantity and quality | Baseline to week 10.
  Change in sleep quantity and quality to be measured via change in total sleep time (TST) and waking after sleep onset (WASO) via the use of wearables.
The impact of CARDIO capsules on cough symptoms from baseline to end of study | Baseline to week 10
  VAS score will be used to assess cough over the preceding 24 hours, measured each morning, on a 100mm scale. The VAS is easy and simple to complete and has been shown to be highly responsive to change in cough symptoms

SECONDARY OUTCOMES:
Subjective Sleep Quality | Baseline to 8 weeks
  Subjective assessment of sleep quality via 100mm VAS with 0mm representing the "best possible sleep" and 100mm representing the "worst possible sleep".
Pro- and Anti-Inflammatory Gene Expression | Baseline to 8 weeks
  Change in gene expression of inflammatory and anti-inflammatory genes (CSF2, CXCL8, IL10, TNF, IL6, IL4, IL5, TGFB1, IL13, BMP2, CRP) encoding cytokines and chemokines will be assessed using nasal swab specimens. Quantitative real-time PCR (qRT-PCR) with TaqMan probe technology will be utilized to measure gene expression levels. This analysis is voluntary and will be conducted in up to 40 subjects.

OTHER OUTCOMES:
Correlation Between AQI and Cough Severity | Baseline to 8 weeks
  Explore the potential correlation between AQI (numerical index on standardized scale) in participants' neighborhoods and cough severity (on a 100-mm linear scale ranging from "no cough" [0 mm] to "worst cough" [100 mm] ) during the intervention period. Correlation will be assessed using Pearson correlation coefficient.

CONTACTS AND LOCATIONS:
Locations (1):
- Alethios, Inc., San Francisco, California, United States

IPD SHARING:
Plan to Share IPD: No